CLINICAL TRIAL: NCT00730067
Title: Sildenafil for COPD-associated Pulmonary Hypertension. A Randomized Double Blinded Placebo Controlled Study.
Brief Title: Sildenafil for Chronic Obstructive Pulmonary Disease (COPD) Associated Pulmonary Hypertension
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: As a single center, it was not possible to recruit enough patients with pulmonary hypertension
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Andersen, MD, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-002237-73
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: COPD; Pulmonary Hypertension
Keywords: COPD; Pulmonary hypertension; Sildenafil; NT-pro BNP; apelin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Sildenafil treatment
  Interventions: Drug: sildenafil
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sildenafil — Sildenafil 50 mg three times daily
  Other Names: Viagra
  Arms: 1
Drug: placebo — tablet with Laetose mono hydrat, talc,Potato tarch, Gelatin, Magnesium stearate.
  Arms: 2

SUMMARY:
Chronic obstructive pulmonary disease (COPD)can be complicated by an increased pressure in the pulmonary circulation. This worsens the prognosis, but so far it is unknown whether treatment of the increased pulmonary blood pressure betters the patients symptoms.

In this study 32 patients with increased pulmonary blood pressure due to COPD will be randomized to 3 months treatment with placebo or sildenafil, which is known to lower the pulmonary blood pressure in other types of pulmonary hypertension.

Our hypothesis is that treatment with sildenafil in these patients will improve the functional capacity measured by the distance walked in 6 minutes and life quality.

ELIGIBILITY:
Inclusion Criteria:

* A mean pulmonary arterial pressure of 25 mmHg measured by right heart catheterization.
* A diagnosis of COPD-associated pulmonary hypertension, implicating that no other potential cause of pulmonary hypertension is present.
* Stable COPD, defined by no subjective alterations of symptoms or use of short acting beta-antagonists for minimally six weeks. Any exacerbation resulting in admission to hospital or other contacts to a physician must have ceased for at least 6 weeks before entering the study.
* Age > 18
* Informed written consent.
* Reliable anticonception for fertile women.

Exclusion Criteria:

* Rheumatic disease limiting walking capacity.
* Exacerbation in COPD during the study.
* Age>80 years
* FEV1 < 25 % of predicted.
* Allergy towards contents of sildenafil or placebo tablets.
* Fall in blood pressure of > 30 mmHg systolic or >20 mmHg diastolic after intake of the first dose of trial medication.
* Fall in peripheral saturation of > 5% after intake of the first dose of trial medication.
* Treatment with nitrous vasodilators or aminophyllamines.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test | at base line, after 2 hours and after 3 months

SECONDARY OUTCOMES:
assessment of life quality | At baseline and follow up after three months
Systolic pulmonary pressure | At baseline and follow-up after three months
Activity of symptoms measured by use of short acting beta agonists | At baseline and follow-up after three months
Levels of NT-proBNP and apelin | At baseline and follow-up after three months

CONTACTS AND LOCATIONS:
Overall Officials: Ole Hilberg, MDSC, Principal Investigator — Århus Sygehus; Jens Erik Nielsen-Kudsk, MDSC, Principal Investigator — Skejby Sygehus
Locations (2):
- Denmark (2):
  - Department of Pulmonary Diseases, Århus Sygehus, Aarhus
  - Department of Cardiology, Skejby sygehus, Århus N